CLINICAL TRIAL: NCT02780804
Title: A Phase 1 Study of Entinostat, an Oral Histone Deacetylase Inhibitor, in Pediatric Patients With Recurrent or Refractory Solid Tumors, Including CNS Tumors and Lymphoma
Brief Title: Entinostat in Treating Pediatric Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-00708; NCI-2016-00708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1513; ADVL1513 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1513 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2016-05-23; First posted 2016-05-24 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Brain Stem Neoplasm; Pineal Region Neoplasm; Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Primary Central Nervous System Neoplasm; Recurrent Visual Pathway Glioma; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm; Refractory Visual Pathway Glioma
MeSH Terms: conditions — Brain Stem Neoplasms; Pinealoma; Lymphoma; Central Nervous System Neoplasms | interventions — entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (entinostat) (Experimental): Patients receive entinostat PO on days 1, 8, 15, and 22. Cycles repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entinostat; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Entinostat — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of entinostat in treating pediatric patients with solid tumors that have come back or have not responded to treatment. Entinostat may block some of the enzymes needed for cell division and it may help to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of entinostat administered as a single-agent, once weekly to children with recurrent or refractory solid tumors.

II. To define and describe the toxicities of entinostat administered as a single agent, once weekly to children with recurrent or refractory solid tumors.

III. To characterize the pharmacokinetics of entinostat in children with recurrent or refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of entinostat within the confines of a phase 1 study.

II. To assess change in histone H3 and H4 acetylation in peripheral blood mononuclear cells (PBMCs) as a marker of the biologic activity of entinostat.

OUTLINE: This is a dose escalation study.

Patients receive entinostat orally (PO) on days 1, 8, 15, and 22. Cycles repeat every 28 days for up to 5 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area (BSA) of >= 1.17 m^2 at time of study enrollment
* Patients must be able to swallow intact tablets
* Patients with recurrent or refractory solid tumors, including central nervous system (CNS) tumors or lymphoma, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; Note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the defined eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

    * Solid tumor patients: >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
    * Lymphoma patients:

      * a waiting period prior to enrollment is not required for patients receiving standard cytotoxic maintenance chemotherapy (i.e. corticosteroid, vincristine, thioguanine[6MP], and/or methotrexate)
      * >=14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea, for patients not receiving standard maintenance therapy; additionally, patients must have fully recovered from all acute toxic effects of prior therapy; Note: cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days must have elapsed from the last dose of agent; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Hematopoietic growth factors: >= 14 days must have elapsed from the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days must have elapsed from the last dose of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without traumatic brain injury [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days must have elapsed from infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days must have elapsed from infusion
  * Cellular therapy: >= 42 days must have elapsed from last dose of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * External beam radiation (XRT)/external beam irradiation including protons: >= 14 days must have elapsed after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, iobenguane I-131 [131I-MIBG]): >= 42 days must have elapsed from the last dose of systemically administered radiopharmaceutical therapy
  * Histone deacetylase (HDAC) inhibitors: Patients must not have received prior therapy with entinostat; patients who have received therapy with other HDAC inhibitors are eligible
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment)
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (within 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dl, with or without transfusion (within 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will not be eligible
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6 mg/dL for males and females
  * 2 to < 6 years: 0.8 mg/dL for males and females
  * 6 to < 10 years: 1.0 mg/dL for males and females
  * 10 to < 13 years: 1.2 mg/dL for males and females
  * 13 to < 16 years: 1.5 mg/dL for males and 1.4 mg/dL for females
  * > = 16 years: 1.7 mg/dL for males and 1.4 mg/dL for females (within 7 days prior to enrollment)
* Bilirubin (sum of conjugated + conjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x upper limit of normal (ULN) = 135 U/l; for the purpose of this study, the ULN for SGPT is 45 U/l (within 7 days prior to enrollment)
* Serum albumin >= 2 g/dl (within 7 days prior to enrollment)
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method both during and for 3 months after participation in this study; abstinence is an acceptable method of contraception; those who become pregnant while on treatment with entinostat must discontinue immediately and consult their treating physician
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients requiring concurrent administration of valproic acid are not eligible for this trial
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients with a BSA ˂ 1.17 m^2 at time of study enrollment are not eligible
* Patients who are not able to swallow intact tablets are not eligible
* Patients with a known history of corrected QT (QTc) prolongation (> 480 msec), or known history of ventricular tachycardia, ventricular fibrillation or Torsades de pointes are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with a history of allergy to medications that have a benzamide structure (e.g., metoclopramide, procarbazine, domperidone, cisapride etc.) are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bukowinski, Principal Investigator — COG Phase I Consortium
Locations (21):
- United States (21):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1 With 3 mg/m²: Patients with recurrent or refractory solid tumors, including lymphoma and CSN tumors, treated once weekly with entinostat administered as a single-agent at 3 mg/m2
- Stratum 1 With 4 mg/m²: Patients with recurrent or refractory solid tumors, including lymphoma and CSN tumors, treated once weekly with entinostat administered as a single-agent at 4 mg/m2
- PK Part With 4 mg/m²: Patients with recurrent or refractory solid tumors without bone marrow involvement, including lymphoma and CSN tumors, treated once weekly with entinostat administered as a single-agent at the RP2D (4 mg/m2)
Period: Overall Study
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Started | 6 | 9 | 6
Completed | 0 | 0 | 0
Not Completed | 6 | 9 | 6
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 8 | 4
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m² | Total
Number analyzed (Participants) | 6 | 9 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants] — Patients must be ≥ than 12 months and ≤ 21 years of age at the time of study enrollment, and Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age.
  Participants
    <=18 years | 4 | 9 | 5 | 18
    Between 18 and 65 years | 2 | 0 | 1 | 3
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 17.5 [13 to 20] | 13 [8 to 17] | 11 [6 to 19] | 14 [6 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 11
  Male | 4 | 4 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 5 | 6 | 5 | 16
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 6 | 6 | 3 | 15
  More than one race | 0 | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (R2PD) of Entinostat
Description: The MTD/RP2D will be defined as the maximum dose at which fewer than one-third of patients experience dose limiting toxicity during cycle 1 of therapy among 6 toxicity-evaluable patients. The frequency of cycle 1 dose limiting toxicities will be summarized by dose level among patients in the dose escalation part of the study.
Time Frame: Up to 28 days
Measure: Number; unit: mg/m²
Groups:
- Treatment (Entinostat): Patients with recurrent or refractory solid tumors, including lymphoma and CNS tumors, who receive entinostat on Days 1, 8, 15, and 22 of a 28-day cycle
Arm/Group | Treatment (Entinostat)
Number analyzed (Participants) | 21
mg/m² | 4

2. Primary Outcome: Frequency of Adverse Events for Entinostat
Description: The frequency of patients with at least one Grade 3 or greater adverse event that are at least possibly attributable to entinostat during cycle 1 will be summarized by study part, dose level.
Time Frame: Up to 28 days
Population: All eligible enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
Participants | 5 | 7 | 5

3. Primary Outcome: Half-life of Entinostat
Description: The median (min, max) Half-Life of entinostat stratified by study part and dose level. The half-life (t1/2) was calculated using the equation t1/2 = 0.693/λz, where the terminal elimination rate constant (λz) was determined from a least-squares regression of the log-transformed plasma concentration vs. time data for the last 3 - 4 time points.
Time Frame: Plasma concentrations were measured at 0, 0.5, 1, 3, 6, 24, and 48-96 hours post-dose during cycle 1, day 1.
Population: All eligible enrolled patients.
Measure: Median (Full Range); unit: Hours
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
Hours | 50.96 [27.38 to 103.66] | 46.04 [40.51 to 81.32] | 44.23 [29.86 to 103.74]

4. Primary Outcome: Peak Plasma Concentration of Entinostat: C-Max
Description: The median (min, max) of the peak plasma concentration of entinostat stratified by study part, dose level. Time points were assessed at 0, 0.5, 1, 3, 6, 24, and 48-96 hours post-dose during cycle 1, day 1.
Time Frame: Up to 96 hours
Population: All eligible enrolled patients.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
ng/ml | 54.4 [5.19 to 136.00] | 61.5 [14.00 to 107.00] | 23.8 [19.10 to 293.00]

5. Primary Outcome: Total Area Under the Plasma Concentration Curve of Entinostat: AUC
Description: The median (min, max) of the total area under the plasma concentration curve of entinostat stratified by study part, dose level. Time points were assessed at 0, 0.5, 1, 3, 6, 24, and 48-96 hours post-dose during cycle 1, day 1.
Time Frame: Up to 96 hours
Population: All eligible enrolled patients.
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
hr*ng/mL | 755 [252 to 1320] | 1111 [816 to 1910] | 1147 [1074 to 2349]

6. Primary Outcome: Time to Reach Maximum Plasma Concentration of Entinostat: T-Max
Description: The median (min, max) of the time to reach maximum plasma concentration of entinostat stratified by study part, dose level. Time points were assessed at 0, 0.5, 1, 3, 6, 24, and 48-96 hours post-dose during cycle 1, day 1.
Time Frame: Up to 96 hours
Population: All eligible enrolled patients.
Measure: Median (Full Range); unit: Hours
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
Hours | 1.01 [0.53 to 6.00] | 0.59 [0.50 to 24.55] | 1 [0.50 to 24.08]

7. Secondary Outcome: Antitumor Activity of Entinostat
Description: Frequency of response to entinostat per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and/or assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR, stratified by study part and dose
Time Frame: Up to 4 years 9 months
Population: All eligible enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 6 | 9 | 6
Participants | 0 | 0 | 0

8. Secondary Outcome: Change in Histone H3 Acetylation of Entinostat
Description: Median (IQR) change in H3 acetylation in peripheral blood mononuclear cells (PBMCs) versus baseline stratified by study part, dose level.
Time Frame: Up to 28 days
Population: Data were not collected
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Histone H4 Acetylation of Entinostat
Description: Median (IQR) change in H4 acetylation in PBMCs versus baseline stratified by study part, dose level.
Time Frame: Up to 28 days
Population: Data were not collected
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years 9 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Stratum 1 With 3 mg/m² | Stratum 1 With 4 mg/m² | PK Part With 4 mg/m²
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/9 | 2/6
Serious Adverse Events (participants affected / at risk) | 5/6 | 7/9 | 5/6
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 3 mg/m² (N=6) | Stratum 1 With 4 mg/m² (N=9) | PK Part With 4 mg/m² (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abducens nerve disorder (Nervous system disorders) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Delusions (Psychiatric disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Eye disorders - Other, HEMIANOPSIA/FIELD CUT (Eye disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 3 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 With 3 mg/m² (N=6) | Stratum 1 With 4 mg/m² (N=9) | PK Part With 4 mg/m² (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2
Abducens nerve disorder (Nervous system disorders) | 1 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 6 | 3
Alkaline phosphatase increased (Investigations) | 1 | 3 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 1
Anxiety (Psychiatric disorders) | 4 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 7 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 2 | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Blood and lymphatic system disorders - Other, ANC INCREASED (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 1 | 1
Blurred vision (Eye disorders) | 3 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Creatinine increased (Investigations) | 2 | 3 | 0
Cushingoid (Endocrine disorders) | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Delusions (Psychiatric disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2
Dry eye (Eye disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Ear and labyrinth disorders - Other, EAR BLEEDS (Ear and labyrinth disorders) | 0 | 0 | 1
Ear and labyrinth disorders - Other, NOISE SENSITIVITY (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Edema face (General disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 2 | 2 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Endocrine disorders - Other, POLYDIPSIA (Endocrine disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Eye disorders - Other, LEFT EYE PROPTOSIS (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, VISUAL FIELD DEFICIT (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, subconjunctival hemorrhage, bilateral (Eye disorders) | 1 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 2
Facial nerve disorder (Nervous system disorders) | 3 | 1 | 0
Facial pain (General disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fatigue (General disorders) | 3 | 6 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 1 | 0
Fever (General disorders) | 2 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal disorders - Other, HEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, INCREASED SALIVARY OUTPUT (Gastrointestinal disorders) | 1 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 5 | 4 | 3
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 1 | 2
Hemoglobin increased (Investigations) | 1 | 3 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 6 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 4 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 3 | 2
Hypoglossal nerve disorder (Nervous system disorders) | 2 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 5 | 4
Hypotension (Vascular disorders) | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1
IVth nerve disorder (Nervous system disorders) | 1 | 0 | 0
Infections and infestations - Other, bicarbonate level increased (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, right hip laceration (Infections and infestations) | 1 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 1
Injury, poisoning and procedural complications - Other, Cut (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, HIT HEAD ON WALL (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, KNEE INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, LIP INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, LOWER EYE LID TISSUE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, SKIN EXORIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poisoning and procedural complications - Other, facial laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 1
Investigations - Other, ALKALINE PHOSPHATASE DECREASED (Investigations) | 0 | 1 | 0
Investigations - Other, BICARB DECREASED (Investigations) | 1 | 0 | 0
Investigations - Other, BICARBONATE DECREASED (Investigations) | 0 | 1 | 0
Investigations - Other, BICARBONATE LEVEL ELEVATED (Investigations) | 1 | 0 | 0
Investigations - Other, BUN ELEVATED (Investigations) | 1 | 0 | 0
Investigations - Other, BUN LOW (Investigations) | 1 | 0 | 0
Investigations - Other, D-DIMER INCREASED (Investigations) | 0 | 0 | 1
Investigations - Other, ELEVATED BUN (Investigations) | 1 | 0 | 1
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 0 | 2
Investigations - Other, Elevated BUN (Investigations) | 0 | 0 | 1
Investigations - Other, FIBRINOGEN INCREASED (Investigations) | 0 | 0 | 1
Investigations - Other, HYPERAMMONEMIA (Investigations) | 0 | 1 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 0 | 2
Investigations - Other, INCREASED PROTHROMBIN TIME (Investigations) | 1 | 0 | 0
Investigations - Other, LACTATE ELEVATED (Investigations) | 0 | 1 | 0
Investigations - Other, LOW BICARB (Investigations) | 0 | 0 | 1
Investigations - Other, LOW BICARBONATE (Investigations) | 0 | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 4 | 1
Malaise (General disorders) | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 3 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Metabolism and nutrition disorders - Other, ELEVATED PHOSPHROUS (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other, HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other, LOW BICARBONATE (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolism and nutrition disorders - Other, VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, Extremity atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nervous system disorders - Other, ABNORMAL BALANCE (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, HYPOTONIA (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other, PATTERNS OF PARALYSIS: ON THE LEFT, HEMIPLEGIA (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, TROUBLE WITH PROCESSING INFORMATION (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 2 | 2
Nystagmus (Nervous system disorders) | 1 | 1 | 1
Oculomotor nerve disorder (Nervous system disorders) | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pain (General disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 1
Platelet count decreased (Investigations) | 4 | 5 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Psychiatric disorders - Other, ADHD (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders - Other, SLEEP WALKING (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders - Other, skin picking disorder (Psychiatric disorders) | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1 | 0
Reproductive system and breast disorders - Other, TESTICULAR HYDROCELE & SPERMATIC CORD/VARICOCELE (Reproductive system and breast disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0
Serum amylase increased (Investigations) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 4 | 1
Skin and subcutaneous tissue disorders - Other, ABRAISON (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ABRASION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Laceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Laceration, left hip (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, POSSIBE ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SORE ON RIGHT FOREARM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, STRIAE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, TEAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, laceration, finger and foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, laceration, left leg (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, skin tear (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Vascular disorders - Other, AV THROMBUS (Vascular disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 7 | 5
Weight gain (Investigations) | 1 | 0 | 1
Weight loss (Investigations) | 1 | 3 | 0
White blood cell decreased (Investigations) | 4 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT02780804/Prot_SAP_000.pdf